CLINICAL TRIAL: NCT05565144
Title: Brain Hemorrhage on 24h-CT and Functional Outcome in Stroke Patients With Cerebral Amyloid Angiopathy Features on Pre-thrombolysis MRI Treated With Intravenous Thrombolysis
Brief Title: Brain Hemorrhage and Functional Outcome in Stroke Patients With CAA Features on Pre-thrombolysis MRI Treated With Intravenous Thrombolysis (Thrombolysis in CAA) ( Thromb in CAA )
Acronym: Thromb in CAA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2022/DR-03
Record Dates: First submitted 2022-09-23; First posted 2022-10-04 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hemorrhage; Cerebral Amyloid Angiopathy; Stroke
Keywords: functional outcome
MeSH Terms: conditions — Hemorrhage; Cerebral Amyloid Angiopathy; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cerebral amyloid angiopathy (CAA): Patients with CAA treated with intravenous thrombolysis
  Interventions: Other: None, pure observational study

INTERVENTIONS:
Other: None, pure observational study — None, pure observational study

SUMMARY:
Background: In stroke patients treated with intravenous thrombolysis (IVT), presence and high number of strictly lobar cerebral microbleeds (compatible with cerebral amyloid angiopathy, CAA) seems to be associated with increased risk of hemorrhagic transformation, symptomatic hemorrhagic transformation, remote hemorrhage, and poor functional outcome. Some of these reported CAA patients with cerebral microbleeds also had chronic lobar intracerebral haemorrhage. Few data is available on IVT-treated CAA patients showing cortical superficial siderosis. There are no reports studying factors associated with brain hemorrhagic complication or functional outcome inside a group of IVT-treated CAA patients. Our aim was to evaluate brain hemorrhagic complications on 24h-CT and functional outcome after IVT in stroke patients with CAA features on pre-IVT MRI.

Methods: In our stroke center, IVT decision in patients with CAA MRI features is left at the discretion of the treating physician. We retrospectively screened pre-IVT imaging of 959 consecutive IVT-treated stroke patients (between January 2015 and July 2022) without ongoing anticoagulation therapy for probable CAA MRI features defined by modified Boston criteria. After exclusion of 119 patients with lacking MRI (n=47), with MRI showing motion artefacts (n=49) or with alternative chronic brain hemorrhage cause on MRI (n=23), 15 IVT-treated patients with probable CAA on pre-IVT MRI were identified. In these 15 patients, clinical, biological and MRI characteristics were compared between patients with vs. without post-IVT hemorrhage and between patients with poor (MRS 3-6) vs. good (MRS 0-2) functional outcome at discharge.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive IVT-treated stroke patients without ongoing anticoagulation therapy registered in our stroke database presenting probable CAA on pre-IVT MRI
* Patient taken in charge at the CHU of Nîmes between January 2015 and July 2022

Exclusion Criteria:

* patients with ongoing anticoagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive IVT-treated stroke patientswith CAA features (strictly lobar CMB, CSS, or chronic lobar ICH) on pre-treatment MRI therapy registered in our stroke database between January 2015 and July 2022
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-10-02 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
brain hemorrhage | 24 hours after intravenous thrombolysis (IVT)
  brain hemorrhage on non-enhanced CT at 24 hours after IVT (Yes/No)
functional outcome | Up to 3 months. From date of symptom onset until date of hospital discharge, assessed up to 3 months.
  functional outcome at hospital discharge according to the modified Rankin scale (Poor/Good)

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France

REFERENCES:
- [Result] Leonte A, Laurent-Chabalier S, Wacongne A, Parvu T, Hackius M, Thouvenot E, Renard D. Brain hemorrhage on 24h-CT and functional outcome in stroke patients with cerebral amyloid angiopathy features on pre-thrombolysis MRI treated with intravenous thrombolysis: A case series. J Stroke Cerebrovasc Dis. 2023 Feb;32(2):106907. doi: 10.1016/j.jstrokecerebrovasdis.2022.106907. Epub 2022 Nov 25. PMID 36442282